CLINICAL TRIAL: NCT00347295
Title: A Randomised, Double-blinded, Double-dummy, Multi-center, Paralleled Study to Investigate the Safety and Efficacy of Brotizolam (Lendormin) Compared With Estazolam in Insomnia Outpatients.
Brief Title: Randomised, Double-blind Study to Investigate the Safety and Efficacy of Brotizolam in Insomnia Outpatients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 263.510
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — brotizolam; Estazolam

INTERVENTIONS:
Drug: Brotizolam
Drug: Estazolam

SUMMARY:
To investigate the efficacy and safety of Brotizolam in the treatment of patients with insomnia in comparison with that of Estazolam

DETAILED DESCRIPTION:
It is intended to recruit 240 insomnia outpatients in this study, 120 patients receiving Brotizolam + Estazolam placebo (Test Group) and 120 patients given Estazolam + Brotizolam placebo (Control Group).

Study Hypothesis:

Brotizolam can be safely used in insomnia patients in China. And Brotizolam 0.25mg is non-inferior with Estazolam 1-2mg in treatment of insomnia patients in China

Comparison(s):

Estazolam 1-2mg

ELIGIBILITY:
Inclusion_Criteria:

Patients will be eligible for enrollment of this study if they meet all of the following criteria:

* Willing and able to provide written informed consent
* Male or female, aged 18 - 65 (including 18 and 65)
* Diagnosed as insomnia by the criteria of CCMD-3:

Exclusion_Criteria:

* Who received any central nervous system drugs within one week before visit 2(baseline)
* Continuous use of hypnotic agents for more than 3 months recently
* History of inefficiency with benzodiazepine-type hypnotics
* Who have a history of obvious hypersensitivity
* Hamilton Depression Rating Scale (HAMD)18
* Who was diagnosed with other mental illness
* With serious diseases of heart, liver and kidney, etc
* Who had sleep apnoea syndrome
* Who had epileptic seizures within one year
* With angle closure glaucoma that is acute or easy to occurred
* Whose AST or ALT values are 2 times of normal upper limit
* Whose Cr or BUN values are 2 times of normal upper limit
* Who are known to be prone to the abuse of alcohol (i.e. history of evidence of acute or chronic abuse), or any other addictive agents
* Who is participating in other clinical trial, or have participated in a clinical study of any other drug in one month prior to visit 2 (baseline). In addition, patients who has been randomized in this trial and then withdrew can not be enrolled again.
* All pregnant, lactational women and women who have the plan of pregnancy.
* Who are unwilling to or not able to complete the whole clinical trial
* Other patients who are unsuitable to be included in the trial judged by investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253
Dates: Start 2006-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01

PRIMARY OUTCOMES:
change of Sleeping Dysfunction Rating Scale (SDRS) total score of Brotizolam in comparison with Estazolam after a 14-day oral administration in patients with insomnia.

SECONDARY OUTCOMES:
The Clinical Global Impression- Improvement score(CGI-I) The Clinical Global Impression- Severity score (CGI-S) Effective rate Rebound phenomena

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (8):
- China (8):
  - Third Hospital of Beijing Hospital, Beijing
  - Beijing Anding Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Guanzhou Psychiatric Hospital, Guangzhou
  - Shanghai Mental Health Center, Shanghai
  - Hu Shan Hospital, Fu Dan University, Shanghai
  - Tongji Hospital, Tongji University, Shanghai

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/23025837